CLINICAL TRIAL: NCT04821687
Title: A Randomized, Parallel Group, Multicenter, Prospective, Open-label, Exploratory, Phase 4 Study to Evaluate the Add-on Effect of Opicapone 50 mg or Levodopa 100 mg as First Strategy for the Treatment of Wearing-off in Patients With Parkinson's Disease
Brief Title: A Study to Evaluate the add-on Efficacy and Safety of Opicapone 50 mg or an Extra Dose of L-DOPA 100 mg for the Treatment of Wearing-off in Patients With PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGT001
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: COMT inhibitor
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opicapone 50mg (Experimental)
  Interventions: Drug: Ongentys 50mg
- Levodopa 100mg (Active Comparator)
  Interventions: Drug: Madopar Tab. 125 or Perkin Tab. 25-100mg

INTERVENTIONS:
Drug: Ongentys 50mg — Opicapone 50mg will be added to current and stable therapy of L-DOPA/DDCI
  Arms: Opicapone 50mg
Drug: Madopar Tab. 125 or Perkin Tab. 25-100mg — Madopar Tab. 125 or Perkin Tab. 25-100mg will be added to current and stable therapy of L-DOPA/DDCI
  Arms: Levodopa 100mg

SUMMARY:
A Study to evaluate the add-on efficacy and safety of opicapone 50 mg or an extra dose of L-DOPA 100 mg for the treatment of wearing-off in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (2006) or according to the Movement Disorder Society (MDS) Clinical Diagnostic Criteria (2015).
2. Disease severity Stage III (H&Y staging) at ON.
3. Treated on a stable regimen for at least four weeks before screening with immediate-release L-DOPA/DDCI, three to four intakes per day, and up to maximum daily dose of 600mg L-DOPA.
4. Signs of wearing-off phenomenon with average total daily OFF-time while awake of at least 1 hour, including the early morning pre-first dose OFF (i.e. the time between wake-up and response to the first L-DOPA/DDCI dosage), despite optimal anti-PD therapy (based on Investigator's assessment).

Exclusion Criteria:

1. Non-idiopathic PD (atypical Parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome.
2. Severe and/or unpredictable OFF periods, according to Investigator judgment.
3. Average total daily OFF-time while awake of >5 hours, including the early morning pre-first dose OFF, despite optimal anti-PD therapy (based on Investigator's assessment).
4. Treatment with prohibited medication: entacapone, tolcapone, monoamine oxidase (MAO) inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation, rasagiline up to 1 mg/day or safinamide up to 100 mg/day), apomorphine or antiemetics with antidopaminergic action (except domperidone) within the last four weeks before screening.
5. Previous or planned (during the entire study duration) deep brain stimulation or stereotactic surgery (e.g. pallidotomy, thalamotomy).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Hauser's diary | Baseline, at 2 weeks, and 4 weeks
  Change in absolute OFF-time and ON-time. Since this study is exploratory, there is no separate primary endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea